CLINICAL TRIAL: NCT05307159
Title: Effect of a Bean (Phaseolus Vulgaris L.) Protein-added Supplement on Body Composition in High-performance Adolescent Athletes: a Pilot Study
Brief Title: Effect of a Bean Protein-added Supplement on Body Composition in High-performance Adolescent Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional de Alta Especialidad de la Península de Yucatán (Other)
Responsible Party: Principal Investigator, Azalia Avila Nava, PhD, Principal Investigator, Hospital Regional de Alta Especialidad de la Península de Yucatán
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-005
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-06

CONDITIONS: Teenagers; Athletes
Keywords: teenagers; bean; supplement; muscle mass; sporty
MeSH Terms: conditions — Spinocerebellar Ataxia 31

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bean protein supplement (Experimental): The supplement will be consumed daily for 21 days in the athletes' snack, the supplement contains 7 g of bean protein mixed in 60 mL of milk and 60 mL of strawberry drinkable yogurt
  Interventions: Dietary Supplement: bean protein supplement

INTERVENTIONS:
Dietary Supplement: bean protein supplement — They will have a snack with bean protein for 21 days Participants will follow their usual diet, which will be quantified and evaluated.

SUMMARY:
Background: Sport is a specialized competitive physical activity that is regulated and requires daily physical training. The workouts allow athletes to increase strength, endurance exercise performance, and muscle mass. Due to this, it is extremely important to consider that high-performance athletes require a meal plan with a higher energy requirement compared to a normal person who does not perform high-intensity activity. The diet of these athletes needs higher protein requirements to support the accumulation and/or maintenance of lean mass. Specifically athletes between 4 to 17 years of age, the protein requirement is of utmost importance to maintain muscle mass between 68-73%. Therefore, the recommendations for protein intake for athletes in this age range is approximately between 10 and 30% of the total energy intake. One of the strategies that has been used is supplementation with protein isolates, since in this way there is greater protein accessibility to maintain a balance between protein synthesis and degradation. The main protein supplements that are currently consumed come from proteins of animal origin; however, these usually have high costs, which makes them difficult to access for the population. Due to this, strategies have begun to be sought through the use of different proteins to generate similar effects.

Objective: To evaluate the effect of a bean protein supplement on body composition in high-performance adolescent athletes.

Methodology: The protocol will be divided into two stages, in the first one a supplement added with bean protein will be elaborated. First, the extraction of protein from the bean will be carried out, then it will be subjected to a heat treatment to eliminate anti-nutrients and finally its chemical composition will be analyzed. In the second stage, a pilot study will be carried out to evaluate the effect of the bean protein supplement in high-performance adolescent athletes. High-performance table tennis athletes, adolescents who agree to collaborate with the study will be included. Bean protein supplementation will be for 21 continuous days in the athletes' snack. Anthropometric measurements will be taken at the beginning and at the end of the intervention. A control of the diet and supplementation of the athletes will be carried out with the support of their coaches.

DETAILED DESCRIPTION:
The protocol will include high-performance table tennis athletes, adolescents who are a minimum of 11 years old and a maximum of 18 years and 11 months who have the consent of their parents and/or guardians and the assent signed by them. Bean protein supplementation will be a mesocycle of 21 continuous days. The supplement will be consumed daily during these 21 days in the athletes' snack. Anthropometric measurements will be taken at the beginning and at the end of the intervention. Their usual diet and adherence to the supplementation of the athletes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Athletes who play table tennis
* Age between 11 and 18 years
* Male and female
* Signature of informed consent by parents or guardians
* Approval of the informed assent by the minor under 18 years of age

Exclusion Criteria:

* High-performance athletes who are injured
* Athletes who are not carrying out a quantified diet
* Athletes who present any pathology and/or consume any medication
* Athlete who consumes another nutritional supplement

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Kilograms of muscle mass | 21 days
  Muscle tissue in relation to total body weight and is estimated from body folds

SECONDARY OUTCOMES:
Percentage of fat Mass | 21 days
  Fat mass is determined through panicle measurements using the ISAK method.
Kilograms of body weight | 21 days
  Measured in kilograms, using the scale

CONTACTS AND LOCATIONS:
Overall Officials: Azalia Ávila-Nava, Principal Investigator — Hospital Regional de Alta Especialidad de la Península de Yucatán
Locations (1):
- Hospital Regional de Alta Especialidad de la Península de Yucatán, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nemet D, Eliakim A. Pediatric sports nutrition: an update. Curr Opin Clin Nutr Metab Care. 2009 May;12(3):304-9. doi: 10.1097/MCO.0b013e32832a215b. PMID 19337125
- [Background] Shenoy S, Dhawan M, Singh Sandhu J. Four Weeks of Supplementation With Isolated Soy Protein Attenuates Exercise-Induced Muscle Damage and Enhances Muscle Recovery in Well Trained Athletes: A Randomized Trial. Asian J Sports Med. 2016 May 23;7(3):e33528. doi: 10.5812/asjsm.33528. eCollection 2016 Sep. PMID 27826398
- [Background] Tang JE, Moore DR, Kujbida GW, Tarnopolsky MA, Phillips SM. Ingestion of whey hydrolysate, casein, or soy protein isolate: effects on mixed muscle protein synthesis at rest and following resistance exercise in young men. J Appl Physiol (1985). 2009 Sep;107(3):987-92. doi: 10.1152/japplphysiol.00076.2009. Epub 2009 Jul 9. PMID 19589961
- [Background] Avila-Nava A, Noriega LG, Tovar AR, Granados O, Perez-Cruz C, Pedraza-Chaverri J, Torres N. Food combination based on a pre-hispanic Mexican diet decreases metabolic and cognitive abnormalities and gut microbiota dysbiosis caused by a sucrose-enriched high-fat diet in rats. Mol Nutr Food Res. 2017 Jan;61(1). doi: 10.1002/mnfr.201501023. Epub 2016 Aug 8. PMID 27352915